CLINICAL TRIAL: NCT06201416
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Activity of Single Ascending Doses of SBT777101 in Subjects With Rheumatoid Arthritis
Brief Title: Study of Single Doses of SBT777101 in Subjects With Rheumatoid Arthritis
Acronym: Regulate-RA
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sonoma Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SBT777101-01
Record Dates: First submitted 2024-01-01; First posted 2024-01-11 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; safety; regulatory T cells; CART; Treg; Inflammatory disease; autoimmune disease; autologous; cell therapy
MeSH Terms: conditions — Arthritis, Rheumatoid; Autoimmune Diseases

STUDY DESIGN:
Intervention Model Description: Sequential escalating dose cohorts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- SBT777101 Dose 1 (Experimental): Low dose SBT777101
  Interventions: Biological: SBT777101
- SBT777101 Dose 2 (Experimental): Mid dose SBT777101
  Interventions: Biological: SBT777101
- SBT777101 Dose 3 (Experimental): High dose SBT777101
  Interventions: Biological: SBT777101

INTERVENTIONS:
Biological: SBT777101 — Experimental treatment

SUMMARY:
This study will test the safety and effects of SBT777101 when given as a single dose to subjects with rheumatoid arthritis. It is the first study of this treatment being done in humans. Increasing dose levels will be given after the safety at lower dose levels is shown.

DETAILED DESCRIPTION:
The study evaluates the safety and effects of a novel regulatory CARTreg cell-based autoimmune and inflammatory disease therapy for the treatment of rheumatoid arthritis. The therapy is an autologous (using the patient's own cells) Treg cell therapy that targets proteins in the inflamed, disease-associated tissue, with the aim to dampen inflammation and restore balance to the immune system.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) <35 kg/m^2, inclusive
* Adult-onset, moderate-to-severe rheumatoid arthritis (RA)
* Moderate-to-severe active disease
* Clinical and/or ultrasound evidence of synovitis
* Prior inadequate response to or unable to tolerate available RA therapies
* Stable doses of RA medications for at least 30 days
* Use of highly effective methods of contraception

Exclusion Criteria:

* Major surgery within 12 weeks prior to screening or planned within 12 months after dosing
* Uncontrolled cardiovascular, pulmonary, renal, hepatic, endocrine, or gastrointestinal disease
* Recurrent infections or active infection
* Active or untreated latent tuberculosis
* Primary or secondary immunodeficiency
* History of or current inflammatory joint disease other than RA

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Incidence, nature, and severity of adverse events [Safety and Tolerability] | Day of treatment to end of follow-up period (48 weeks)
Incidence and nature of dose-limiting toxicities (DLTs) | Day of treatment to end of DLT evaluation period (28 days)
  Death, CRS, ICANS, vital organ toxicity, hematological toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Arron, MD, Study Director — Sonoma Biotherapeutics, Inc.
Locations (8):
- United States (8):
  - Mayo Clinic, Scottsdale, Arizona
  - UCSF Medical Center, San Francisco, California
  - Stanford Medical Center, Stanford, California
  - University of Colorado, Aurora, Colorado
  - Northwestern University, Chicago, Illinois
  - Tufts University, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No